CLINICAL TRIAL: NCT04743739
Title: A Multicenter Randomized Controlled Trial of Rituximab Combined With Cyclosporine Versus Rituximab Alone in the Treatment of Idiopathic Membranous Nephropathy
Brief Title: Rituximab Combined With Cyclosporine Versus Rituximab Alone in the Treatment of iMN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient patient enrollment
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); The Luhe Teaching Hospital of the Capital Medical University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iMN RTX plus CsA
Record Dates: First submitted 2021-01-30; First posted 2021-02-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Rituximab; cyclosporine; idiopathic membranous nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab monotherapy (Active Comparator): Rituximab 1000mg I.V. on Days 1 and 181, and will be retreated or not on Days 15 and 195 according to the CD19+ B cells count.
  Interventions: Drug: Rituximab
- Rituximab combined with cyclosporine (Experimental): Rituximab 1000mg I.V. on Days 1 and 181, and will be retreated or not on Days 15 and 195 according to CD19+ B cells count.
  cyclosporine (CsA) will be started at a dose of 3mg/kg/day p.o. divided into 2 equal doses given at 12 hour intervals. Doses of CsA will be adjusted according to the blood levels of CsA. CsA will be tapered after 6 months and discontinued over a 3 month period.
  Interventions: Drug: Rituximab; Drug: cyclosporine

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000mg, I.V. on Days 1 and 181, and will be retreated or not at Days 15 and 195 according to the CD19+ B cell count.
  Other Names: CD20 antibody
Drug: cyclosporine — cyclosporine (CsA) will be started at a dose of 3mg/kg/d and adjusted according to the blood levels of the CsA. CsA will be tapered after 6 months and discontinued over a three month period.
  Other Names: CsA
  Arms: Rituximab combined with cyclosporine

SUMMARY:
The primary objective of this study is to determine whether or not cyclosporine (CsA) combined with RTX is more effective than RTX alone in the treatment of idiopathic membranous nephropathy (iMN).

DETAILED DESCRIPTION:
To date, the first-line immunosuppressive therapy of iMN includes corticosteroids combined with cyclophosphamide or Rituximab (RTX) which has been used more and more widely due to superior safety profiles. But the long term remission rate of RTX monotherapy is only 60% and it takes effect relatively slowly.

2 pilot studies reported that the combination therapy of cyclosporine (CsA) and RTX had better efficacy for inducing remission for iMN, with the long term remission rate up to 85%. CsA and RTX may have synergistic effect in the treatment of iMN because they have different time of action and different effects on the immune system and podocytes.

Based on the previous rationale, the investigators designed this trial to determine whether combination of CsA and RTX is more effective than RTX alone in the treatment of iMN.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic MN with or without diagnostic biopsy
* Female, must be post-menopausal, sterile or have effective method of contraception
* must be off steroid or mycophenolate mofetil for >1 month and alkylating agents for > 6 months
* Angiotensin-converting-enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) for ≥3 months prior to randomization with controlled blood pressure or if patients is intolerant to ACEI/ARB
* proteinuria ≥4g/24h using the average from two 24-hour urine samples collected within 2 weeks of each other, and decreased ≤50% from baseline.
* estimated glomerular filtration rate (eGFR) ≥40ml/min/1.73m2

Exclusion Criteria:

* presence of active infection or a secondary cause of MN
* diabetes mellitus: to exclude proteinuria secondary to diabetic nephropathy.
* pregnancy or breast feeding
* history of resistance to CsA or other calcineurin inhibitors(CNI), RTX or alkylating agents.
* Patients who previously achieved remission after treatment of CNI, RTX or alkylating agents but relapsed off CNI after 3 months, or relapsed off RTX or alkylating agents after 6 months, are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
complete remission (CR) or partial remission (PR) at 24 month | 24 months after randomization
  complete or partial remission at 24 month. complete remission is defined as urine protein≤0.5g/24h and serum albumin≥3.5g/dl. Partial remission is defined as reduction in baseline urine protein ≥50% plus urine protein≤3.5g/24h but >0.5g/24h

SECONDARY OUTCOMES:
complete remission (CR) or partial remission (PR) on 6 month, 12 month, 18 month | 6, 12, 18 months after randomization
  complete or partial remission on month 6, 12 and 18
complete remission (CR) on 6, 12, 18, 24 month | 6, 12, 18, 24 months after randomization
  complete remission on month 6, 12, 18 and 24
Time to complete remission (CR) or partial remission (PR) | from date of randomization until the date of first remission, assessed up to 24 months
  Time to complete or partial remission
Change of estimated glomerular filtration rate (eGFR) | 24 months
  Change of eGFR from baseline to 24 months
Serum creatinine increase≥50 percent from baseline | 24 months
  proportion of patients with increase of serum creatinine ≥50 percent from baseline
Proportion of patients with relapse | 12，18，24 months
  Rate of relapse. Relapse is defined as development of nephrotic range proportion of patients with relapse. Relapse is defined as development of proteinuria>3.5g/24h following CR or PR.
Anti-PLA2R titer | baseline and 3, 6, 9, 12, 18, 24 months
  Auto-antibodies to the M-type phospholipase A2 receptor(PLA2R)
The number of CD19+B cells | baseline and 3, 6, 9, 12, 18, 24 months
  CD19+ B cells
Quality of life measured by kidney disease and quality of life (KDQOL-36) | baseline, 12 and 24 month
  KDQOL-36 includes 36 questions which are scored positively (higher score indicating better quality of life) on a 0-100 scale using developer-recommended scoring.
Adverse events | through study completion until 24 months
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qin, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Tongren Hospital， Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Nanyang Nanshi Hospital, Henan University, Nanyang, Henan
  - The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Shenzhen
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polanco N, Gutierrez E, Covarsi A, Ariza F, Carreno A, Vigil A, Baltar J, Fernandez-Fresnedo G, Martin C, Pons S, Lorenzo D, Bernis C, Arrizabalaga P, Fernandez-Juarez G, Barrio V, Sierra M, Castellanos I, Espinosa M, Rivera F, Oliet A, Fernandez-Vega F, Praga M; Grupo de Estudio de las Enfermedades Glomerulares de la Sociedad Espanola de Nefrologia. Spontaneous remission of nephrotic syndrome in idiopathic membranous nephropathy. J Am Soc Nephrol. 2010 Apr;21(4):697-704. doi: 10.1681/ASN.2009080861. Epub 2010 Jan 28. PMID 20110379
- [Background] Beck LH Jr, Bonegio RG, Lambeau G, Beck DM, Powell DW, Cummins TD, Klein JB, Salant DJ. M-type phospholipase A2 receptor as target antigen in idiopathic membranous nephropathy. N Engl J Med. 2009 Jul 2;361(1):11-21. doi: 10.1056/NEJMoa0810457. PMID 19571279
- [Background] Schreiber SL, Crabtree GR. The mechanism of action of cyclosporin A and FK506. Immunol Today. 1992 Apr;13(4):136-42. doi: 10.1016/0167-5699(92)90111-J. PMID 1374612
- [Background] Faul C, Donnelly M, Merscher-Gomez S, Chang YH, Franz S, Delfgaauw J, Chang JM, Choi HY, Campbell KN, Kim K, Reiser J, Mundel P. The actin cytoskeleton of kidney podocytes is a direct target of the antiproteinuric effect of cyclosporine A. Nat Med. 2008 Sep;14(9):931-8. doi: 10.1038/nm.1857. PMID 18724379
- [Background] Cattran DC, Alexopoulos E, Heering P, Hoyer PF, Johnston A, Meyrier A, Ponticelli C, Saito T, Choukroun G, Nachman P, Praga M, Yoshikawa N. Cyclosporin in idiopathic glomerular disease associated with the nephrotic syndrome : workshop recommendations. Kidney Int. 2007 Dec;72(12):1429-47. doi: 10.1038/sj.ki.5002553. Epub 2007 Sep 26. PMID 17898700
- [Background] Fervenza FC, Appel GB, Barbour SJ, Rovin BH, Lafayette RA, Aslam N, Jefferson JA, Gipson PE, Rizk DV, Sedor JR, Simon JF, McCarthy ET, Brenchley P, Sethi S, Avila-Casado C, Beanlands H, Lieske JC, Philibert D, Li T, Thomas LF, Green DF, Juncos LA, Beara-Lasic L, Blumenthal SS, Sussman AN, Erickson SB, Hladunewich M, Canetta PA, Hebert LA, Leung N, Radhakrishnan J, Reich HN, Parikh SV, Gipson DS, Lee DK, da Costa BR, Juni P, Cattran DC; MENTOR Investigators. Rituximab or Cyclosporine in the Treatment of Membranous Nephropathy. N Engl J Med. 2019 Jul 4;381(1):36-46. doi: 10.1056/NEJMoa1814427. PMID 31269364
- [Background] van den Brand JAJG, Ruggenenti P, Chianca A, Hofstra JM, Perna A, Ruggiero B, Wetzels JFM, Remuzzi G. Safety of Rituximab Compared with Steroids and Cyclophosphamide for Idiopathic Membranous Nephropathy. J Am Soc Nephrol. 2017 Sep;28(9):2729-2737. doi: 10.1681/ASN.2016091022. Epub 2017 May 9. PMID 28487395
- [Background] Segarra A, Praga M, Ramos N, Polanco N, Cargol I, Gutierrez-Solis E, Gomez MR, Montoro B, Camps J. Successful treatment of membranous glomerulonephritis with rituximab in calcineurin inhibitor-dependent patients. Clin J Am Soc Nephrol. 2009 Jun;4(6):1083-8. doi: 10.2215/CJN.06041108. Epub 2009 May 28. PMID 19478097
- [Background] Waldman M, Beck LH Jr, Braun M, Wilkins K, Balow JE, Austin HA 3rd. Membranous nephropathy: Pilot study of a novel regimen combining cyclosporine and Rituximab. Kidney Int Rep. 2016 Jul;1(2):73-84. doi: 10.1016/j.ekir.2016.05.002. Epub 2016 Jun 11. PMID 27942609
- [Background] Fernandez-Juarez G, Rojas-Rivera J, Logt AV, Justino J, Sevillano A, Caravaca-Fontan F, Avila A, Rabasco C, Cabello V, Varela A, Diez M, Martin-Reyes G, Diezhandino MG, Quintana LF, Agraz I, Gomez-Martino JR, Cao M, Rodriguez-Moreno A, Rivas B, Galeano C, Bonet J, Romera A, Shabaka A, Plaisier E, Espinosa M, Egido J, Segarra A, Lambeau G, Ronco P, Wetzels J, Praga M; STARMEN Investigators. The STARMEN trial indicates that alternating treatment with corticosteroids and cyclophosphamide is superior to sequential treatment with tacrolimus and rituximab in primary membranous nephropathy. Kidney Int. 2021 Apr;99(4):986-998. doi: 10.1016/j.kint.2020.10.014. Epub 2020 Nov 7. PMID 33166580